CLINICAL TRIAL: NCT03664037
Title: Dexamethasone Blunts the Hypotensive Effect of Spinal Anesthesia in Geriatric Patients Undergoing Lower Limb Orthopedic Surgeries: a Double Blind, Placebo-controlled Study
Brief Title: Dexamethasone Blunts the Hypotensive Effect of Spinal Anesthesia in Geriatric Patients Undergoing Lower Limb Orthopedic Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor, M.D., Department of Anesthesia and Intensive Care, Ain- shams University, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R 46 / 2018
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D group, (n=55) (Active Comparator)
  Interventions: Drug: Dexamethasone phosphate
- C group, (n=55) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone phosphate — each patient received 8 mg of intravenous DEX diluted in 100 ml 0.9% sodium chloride (normal saline [NS]) intravenous infusion (IVI) over 15 min 2 hours preoperatively
  Arms: D group, (n=55)
Drug: Placebo — each patient received 100 mL 0.9% NS IVI over 15 min (Placebo) 2 hours preoperatively
  Arms: C group, (n=55)

SUMMARY:
Based on the data that DEX increases the TPR and may decrease the expression of serotonin the investigator conducted this study to test the hypothesis that the prophylactic intravenous infusion (IVI) of DEX can attenuate the hypotensive effect of spinal anesthesia in elderly population.

DETAILED DESCRIPTION:
After approval by the institute ethics committee, this study was conducted at Ain-Shams university hospitals, from the 1st of March 2018 till the 31st of August 2018 and on 110 patients aged 60 years or older of the American Society of Anesthesiologists (ASA) physical status I, II or III. A written informed consent was obtained from all patients to participate in the study. Patients with contraindication to SA (e.g. coagulopathy, thrombocytopenia, allergy to local anesthetic agent) and those on steroid or serotonin related medications (e.g. selective serotonin reuptake inhibitor) were excluded.

This study was designed to be a randomized, placebo-controlled, double-blinded parallel study. Following enrollment, patients were randomized into 2 equal groups; the D group, (n=55) each patient received 8 mg of intravenous DEX diluted in 100 ml 0.9% sodium chloride (normal saline [NS]) intravenous infusion (IVI) over 15 min 2 hours preoperatively and the C group, (n=55) each patient received 100 mL 0.9% NS IVI over 15 min (Placebo) 2 hours preoperatively. Randomization was done using computer-generated number table of random numbers in a 1:1 ratio in opaque and sealed envelope (SNOSE). The assigned treatment was written on a card and sealed in opaque envelopes consecutively numbered. These envelopes were opened just immediately before infusing the medication in the patient's room. The study drugs were prepared by the hospital pharmacy and follow-up of patients were conducted by the anesthesia residents not involved in any other part of the study.

Patients were prepared by fasting (8 h for solid foods and 4 hours for clear fluids) before anesthesia and were hydrated intravenously before the procedure. Patients were hooked to a portable monitor (Non-invasive blood pressure and pulse oximetry) in their rooms from which baseline measurements (heart rate(HR), systolic(SAP), diastolic(DAP) and mean arterial blood pressure(MAP)) were recorded just before administration of the study medication.

As soon as the patient arrived in the operating room pulse oximetry, electrocardiogram monitoring, and non-invasive arterial pressure measurement were started, and patients were sedated by 1mg of IV midazolam. An18-gauge intravenous cannula was inserted, and slow infusion of 0.9% sodium chloride solution was commenced to keep the vein opened and didn't exceed the volume of 200 mL during the study period (during giving anesthesia and for 20 minutes thereafter). Lumbar puncture was performed with the patient in a sitting position and the subarachnoid space was punctured at the L3-L4 or L4-L5 level using 25 gauge Quincke spinal needle under aseptic condition. After identification of the subarachnoid space3 mL of 0.5% hyperbaric bupivacaine solution (Marcaine® Spinal 0.5% Heavy; Sunny pivacaine, Manufactured by Sunny Pharmaceutical - Cairo - Egypt) were injected over 60 seconds.

Immediately after completing the subarachnoid injection, patients were positioned supine on the operating table. This was followed by assessment of sensory block every 5 minutes with a cold sensation test (using alcohol swab). At the same time points, the level of motor blockade was assessed (according to the Modiﬁed Bromage Score(13) with the following categories: 0=No motor block; 1=Inability to raise extended leg; able to move knees and feet; 2=Inability to raise extended leg and move knee; able to move feet and 3=Complete block of motor limb), and the HR, SAP, DAP and the MAP were measured and recorded every 5 minutes after SA and for 4 readings thereafter.

Hypotension was considered if there was 25% decrease below the baseline for MAP and was treated with IV crystalloid (Ringer solution) and incremental IV 5 mg doses of ephedrine. Bradycardia was considered if the heart rate < 50 beats/min and was treated with IV atropine (0.01mg/kg).

The study end point was 20 minutes after giving the subarachnoid block during which positioning, raising tourniquet or surgical incision was not be allowed.

Data collection:

The hemodynamic parameter values before anesthesia and the values recorded after the blockade were used for the analysis. Analysis was done by comparing the obtained values at each study time point and by comparing the minimal values recorded within the 20 minutes following the blockade as well. When ephedrine or atropine administration was necessary, only the values obtained before this medication was used. Surgical procedure, positioning the patient or application of tourniquet was not allowed during the study period.

Outcomes:

The primary outcome variable in this study was proportions of patients with hypotension defined as a MAP at least 25% less than the basal value at any time during the first 20 min after induction of SA before start of surgical procedure.

The secondary outcomes were:

* The characteristics of the motor blockade.
* The changes in the MAP, SAP, and DAP values in both patient groups, which were recorded before blockade and at 5-minute intervals after the block (till 20 minutes following the blockade).
* The changes in the heart rate (HR).
* The total ephedrine consumption was given to correct hypotension.
* The total atropine consumption was given to correct bradycardia.

  3-Analysis of Data:

Depending on Baig et al.,2017(14) who found that the hypotension rate in ondansetron and normal saline groups 7.5% and 28.3% respectively, and assuming the power= 0.80 and α=0.05 and by using PASS 11th release the minimal sample size for an equal size controlled clinical trial was 50 in each group. The investigator recruited 55 in each group for possible attrition(15).

The collected data were coded, tabulated, and statistically analyzed using IBM SPSS statistics (Statistical Package for Social Sciences) software version 22.0, IBM Corp., Chicago, USA, 2013.

ELIGIBILITY:
Inclusion Criteria:

* 110 patients aged 60 years or older
* of the American Society of Anesthesiologists (ASA) physical status I, II or III
* undergoing lower limb orthopedic surgeries.
* A written informed consent was obtained from all patients to participate in the study.

Exclusion Criteria:

* Patients with contraindication to SA (e.g.- coagulopathy,
* thrombocytopenia,
* allergy to local anesthetic agent)
* and those on steroid or serotonin related medications (e.g. selective serotonin reuptake inhibitor) were excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
proportions of patients with hypotension defined as a MAP at least 25% less than the basal value at any time during the first 20 min after induction of SA before start of surgical procedure. | The first 20 minutes after induction of SA before start of surgical procedure.
  proportions of patients with hypotension defined as a MAP at least 25% less than the basal value at any time during the first 20 min after induction of SA before start of surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim Mamdouh Esmat, Heliopolis, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Ashoor TM, Hussien NS, Anis SG, Esmat IM. Dexamethasone blunts postspinal hypotension in geriatric patients undergoing orthopedic surgery: a double blind, placebo-controlled study. BMC Anesthesiol. 2021 Jan 11;21(1):11. doi: 10.1186/s12871-021-01232-w. PMID 33430772